CLINICAL TRIAL: NCT05610891
Title: A Phase 1b, Open-Label, Study of a Novel Targeted Radiotherapy in Children, Adolescents and Young Adults With Inoperable Relapsed or Refractory High-Grade Glioma
Brief Title: Novel Targeted Radiotherapy in Pediatric Patients With Inoperable Relapsed or Refractory HGG
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCL-17-001-pHGG; 13460625 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-07

CONDITIONS: High-Grade Glioma
MeSH Terms: conditions — Glioma | interventions — CLR1404

STUDY DESIGN:
Intervention Model Description: Drug: CLR 131 is a radio-iodinated therapy comprising a core phospholipid ether (PLE) analogue radiolabeled with iodine-131. CLR 131 exploits the tumor-targeting properties of PLEs to provide targeted delivery of radiation to malignant tumor cells and minimizes radiation exposure to normal tissues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pediatric High-Grade Glioma Patients (Experimental): Two dosing cohorts will be explored; patients in the first arm will receive two doses, 20 mCi/m2 each, separated by 14 days for two cycles, with a third optional cycle. Patients in the second arm will receive two doses, 10 mCi/m2 each, separated by 14 days for three cycles with a fourth optional cycle.
  Interventions: Drug: CLR 131

INTERVENTIONS:
Drug: CLR 131 — CLR 131 will be administered IV (intravenously) at a dose based on patients' BSA
  Other Names: iopofosine I 131

SUMMARY:
The purpose of this dose finding study is to evaluate the safety and efficacy of 2 different dose levels of CLR 131 in children, adolescents and young adults with relapsed or refractory high-grade glioma (HGG).

DETAILED DESCRIPTION:
This study is designed to further evaluate the safety and tolerability of CLR 131 at the selected doses in children, adolescents and young adults with relapsed or refractory malignant high-grade glioma. It will also determine the therapeutic activity defined as progression free survival and overall survival, antitumor activity (treatment response) defined as the reduction in tumor volume and identify the recommended Phase 2/3 dose of CLR 131 in children, adolescents and young adults with relapsed or refractory HGG.

ELIGIBILITY:
Inclusion Criteria:

* Previously confirmed (histologically or cytologically) high grade glioma that is clinically or radiographically suspected to be relapsed, refractory, or recurrent
* ≥ 10 years of age and ≤ 25 years of age at time of consent/assent
* If ≥ age 16 years, Karnofsky performance status of ≥ 60. If < age 16 years, Lansky performance status ≥ 60
* Platelets ≥ 75,000/μL (last transfusion, if any, must be at least 1 week prior to study registration, and, unless deemed medically necessary, no transfusions are allowed between registration and dosing)
* Absolute neutrophil count ≥ 750/μL
* Hemoglobin ≥ 8 g/dL (last transfusion must be at least 1 week prior to study registration, and, unless deemed medically necessary, no transfusions are allowed between registration and dosing)
* Using the bedside Schwartz formula, estimated GFR (creatinine clearance) > 60 ml/min/1.73m2
* Alanine aminotransferase < 3 × ULN
* Bilirubin < 2 × ULN
* At least 1 measurable intracranial lesion with longest diameter of at least 10 mm on any imaging sequence.
* Patients with previously known neurological deficits must be clinically stable at time of enrollment and able to complete all study related procedures. Patients with documented or newly diagnosed neurological deficits will be enrolled at the investigator's discretion.
* If patient receives steroids for neurological symptom control, the dose must be stable (unchanged for three weeks prior to registration) or on a steroid tapering regimen. Initiation of steroids per routine care immediately prior to CLR 131 dosing is acceptable
* Patient or his or her legal representative is judged by the Investigator to have the initiative and means to be compliant with the protocol.
* Patient or his or her legal representative has the ability to read, understand, and provide written informed consent for the initiation of any study-related procedures.
* Female patients of childbearing potential must have a negative pregnancy test at screening and within 24 hours of dosing. It is recommended that female caregivers of childbearing potential have a negative pregnancy test within one week of dosing.
* Patients of childbearing potential must practice an effective method of birth control while participating on this study to avoid possible harm to the fetus.

Exclusion Criteria:

* Antitumor therapy or investigational therapy, within 3-half-lives of the agent preceding the present study. For certain types of radiation (craniospinal, total abdominal, whole lung [spot irradiation to skull-based metastases is not considered craniospinal radiation for the purposes of this study]), at least 3 months must have elapsed. Palliative focal radiation to non-target lesions should be completed at least 2 weeks prior to dosing. Patients participating in non-interventional clinical trials (i.e., non-drug) are allowed to participate in this trial
* History of hypersensitivity to thyroid protection medication (e.g., potassium iodide, Lugol's solution, etc.)
* Any other concomitant serious illness or organ system dysfunction (including cardiac and pulmonary dysfunction) that in the opinion of the Investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
* Major surgery within 6 weeks of enrollment unless delay in therapy poses unacceptable risk to the patient due to clinical progression (enrollment o such patients should be discussed with Medical Monitor)
* Known history of human immunodeficiency virus or uncontrolled, serious, active infection
* Pregnancy or breast-feeding

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation of CLR 131 | Assessed throughout the study to 1-year post-infusion follow-up period
  Will be assessed by physical examination, performance status, vital signs, laboratory changes over time, and adverse events. Evaluations will use a nonparametric Wilcoxon Signed Rank test and a linear mixed effects modeling will be conducted to evaluate longitudinal changes.
Efficacy Evaluation for Progression Free Survival | Day 84 post-infusion follow-up period through 3 years following completion of treatment.
  To determine the therapeutic activity defined as Progression Free Survival (PFS) using Kaplan Meier estimator. PFS is defined as the time from arm assignment until disease progression or death.

SECONDARY OUTCOMES:
Treatment Response of CLR 131 | From date of arm assignment until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 48 months.
  Determine antitumor activity (treatment response) defined as the reduction in tumor volume, measured by MRI scans acquired as FLAIR images and based on the RAPNO criteria for responses.
Dose Determination for CLR 131 | From date of arm assignment until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 48 months.
  Identify the recommended Phase 2/3 dose of CLR 131 in relapsed pHGG patients based on both safety and efficacy assessments as defined by the primary endpoints concluded from this study.
Dosimetry Evaluation for Total Body and Organ | 4 hours post-infusion and concluding 4 weeks post-initial imaging
  To determine total body and organ dosimetry, together, of CLR 131 in relapsed pHGG patients, measured by conjugate planar whole-body imaging and/or blood collection drawn for radiologic dosimetry analysis for a subset of patients. Organ time/activity integrals will be entered into OLINDA/EXM software to produce total body and organ dosimetry values for CLR 131.
Tumor Response to CLR 131 | 4 hours post-infusion and concluding 4 weeks post-initial imaging
  Determine the tumor uptake of CLR 131 and utility of SPECT/CT as a potential diagnostic for response. Images will be reconstructed using quantitative SPECT reconstruction methods with compensation for attenuation, scatter and the full collimator-detector response including septal penetration and scatter. A registered CT image will be used as the attenuation map for the SPECT images. Image data will be converted to activity per cubic centimeters using a sensitivity measurement made using a point source in air.

CONTACTS AND LOCATIONS:
Overall Officials: Jarrod Longcor, Study Director — Chief Operating Officer
Locations (8):
- United States (7):
  - Stanford University, Palo Alto, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Cancer Center, Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Carbone Cancer Center, Madison, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be made available upon request of NCI, the funding agency partner. This has not yet been decided.